CLINICAL TRIAL: NCT00812357
Title: Descriptive Pharmacoepidemiological Study on the Use of Symbicort Turbuhaler in the Treatment of Asthma in France and Impact of a New Therapeutic Strategy on the Compliance and Control of Asthma
Brief Title: Symbicort Usage in Asthma Treatment and Impact of a New Therapeutic Strategy on Compliance and Asthma Control in France
Acronym: SYMBIOSE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RFR-SYM-2008/1
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Asthma
Keywords: Symbicort Turbuhaler; asthma; cohort study; France
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients treated with Symbicort basic treatment
- 2: Patients treated with Symbicort basic treatment + treatment of symptoms as needed

SUMMARY:
Descriptive pharmacoepidemiological study on the use of Symbicort Turbuhaler in the treatment of asthma in France and impact of a new therapeutic strategy on the compliance and control of asthma

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients treated for this disease with Symbicort Turbuhaler
* Patients monitored for asthma by the doctor for at least 12 months
* Patients seen in outpatient care at the baseline visit
* Patients agreeing to participate in the study

Exclusion Criteria:

* Patients with any chronic lower respiratory disease other than asthma
* Patients receiving anti-IgE agents in the last 4 months
* Patients receiving desensitisation treatment outside of the maintenance phase
* Patients deemed to be unable to respond to the study for linguistic or cognitive reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Level of control of the asthma | 3 months
Evaluation of compliance with treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane SCHÜCK, MD, MSc, Principal Investigator — KAPPA SANTE - Paris - France; Michel AUBIER, MD, Professor, Study Chair — CHU Bichat - Service de pneumologie - Paris - France
Locations (168):
- France (168):
  - Research Site, Dessenheim, Alsace
  - Research Site, Duppigheim, Alsace
  - Research Site, Haguenau, Alsace
  - Research Site, Obernai, Alsace
  - Research Site, Schiltigheim, Alsace
  - Research Site, Strasbourg, Alsace
  - Research Site, Bordeaux, Aquitaine Nord
  - Research Site, Boutiers-Saint-Trojan, Aquitaine Nord
  - Research Site, Bruges, Aquitaine Nord
  - Research Site, Le Bouscat, Aquitaine Nord
  - Research Site, Saujon, Aquitaine Nord
  - Research Site, Hinx, Aquitaine Sud
  - Research Site, Saugnac-et-Cambran, Aquitaine Sud
  - Research Site, Aire-sur-la-Lys, Artois
  - Research Site, Bruay-la-Buissière, Artois
  - Research Site, Marles-les-Mines, Artois
  - Research Site, Ste Austreberthe, Artois
  - Research Site, Aix-en-Othe, Aube Franche Comte
  - Research Site, Belfort, Aube Franche Comte
  - Research Site, Épinal, Aube Franche Comte
  - Research Site, Héricourt, Aube Franche Comte
  - Research Site, Montrond-le-Château, Aube Franche Comte
  - Research Site, Roulans, Aube Franche Comte
  - Research Site, Cournon-d'Auvergne, Auvergne Stephanois
  - Research Site, Le Puy-en-Velay, Auvergne Stephanois
  - Research Site, Pierre-Bénite, Auvergne Stephanois
  - Research Site, Saint-Etienne, Auvergne Stephanois
  - Research Site, Caen, Basse Normandie
  - Research Site, Colleville-Montgomery, Basse Normandie
  - Research Site, Lisieux, Basse Normandie
  - Research Site, Saint-Martin-des-Champs, Basse Normandie
  - Research Site, Dijon, Bourgogne-Franche-Comté
  - Research Site, Fontaine-lès-Dijon, Bourgogne-Franche-Comté
  - Research Site, Le Creusot, Bourgogne-Franche-Comté
  - Research Site, Laval, Bretagne Nord
  - Research Site, Loudéac, Bretagne Nord
  - Research Site, Rennes, Bretagne Nord
  - Research Site, Brest, Bretagne Sud
  - Research Site, Vannes, Bretagne Sud
  - Research Site, Athis-Mons, Brie
  - Research Site, Corbeil-Essonnes, Brie
  - Research Site, Créteil, Brie
  - Research Site, Draveil, Brie
  - Research Site, Férolles-Attilly, Brie
  - Research Site, Yerres, Brie
  - Research Site, Bédarieux, Catalogne
  - Research Site, Béziers, Catalogne
  - Research Site, Bouzigues, Catalogne
  - Research Site, Caunes-Minervois, Catalogne
  - Research Site, Narbonne, Catalogne
  - Research Site, Perpignan, Catalogne
  - Research Site, Saint-André-de-Sangonis, Catalogne
  - Research Site, Sérignan, Catalogne
  - Research Site, Châlons-en-Champagne, Champagne Ardennes
  - Research Site, Reims, Champagne Ardennes
  - Research Site, Châtellerault, Charente
  - Research Site, La Tranche-sur-Mer, Charente
  - Research Site, Niort, Charente
  - Research Site, Poitiers, Charente
  - Research Site, Rochefort, Charente
  - Research Site, Royan, Charente
  - Research Site, Thuré, Charente
  - Research Site, Chambéry, Dauphine
  - Research Site, Grenoble, Dauphine
  - Research Site, La Tronche, Dauphine
  - Research Site, Metz-Tessy, Dauphine
  - Research Site, Saint-Martin-d'Hères, Dauphine
  - Research Site, Antibes, Esterel
  - Research Site, Cagnes-sur-Mer, Esterel
  - Research Site, Draguignan, Esterel
  - Research Site, Le Cannet, Esterel
  - Research Site, Nice, Esterel
  - Research Site, Saint-Laurent-du-Var, Esterel
  - Research Site, Lille, Flandres
  - Research Site, Tourcoing, Flandres
  - Research Site, Douelle, Gascogne
  - Research Site, Lamagistère, Gascogne
  - Research Site, Montauban, Gascogne
  - Research Site, Villeneuve-sur-Lot, Gascogne
  - Research Site, Bois-Guillaume, Haute Normandie
  - Research Site, Pont-de-l'Arche, Haute Normandie
  - Research Site, Rouen, Haute Normandie
  - Research Site, Saint-Saëns, Haute Normandie
  - Research Site, Vernon, Haute Normandie
  - Research Site, Cachan, Hauts de Seine
  - Research Site, Le Kremlin-Bicêtre, Hauts de Seine
  - Research Site, Neuilly-sur-Seine, Hauts de Seine
  - Research Site, Paris, Hauts de Seine
  - Research Site, Arles, Languedoc
  - Research Site, Capdenac-Gare, Languedoc
  - Research Site, Castelnau-le-Lez, Languedoc
  - Research Site, Montpellier, Languedoc
  - Research Site, Rieupeyroux, Languedoc
  - Research Site, Villefranche de Rouergue C, Languedoc
  - Research Site, Ahun, Limousin
  - Research Site, Bourges, Limousin
  - Research Site, Brive-la-Gaillarde, Limousin
  - Research Site, Bruère-Allichamps, Limousin
  - Research Site, Châteauroux, Limousin
  - Research Site, Limoges, Limousin
  - Research Site, Rosiers-d'Égletons, Limousin
  - Research Site, Saint-Yrieix-la-Perche, Limousin
  - Research Site, Forbach, Lorraine
  - Research Site, Metz, Lorraine
  - Research Site, Nancy, Lorraine
  - Research Site, Thionville, Lorraine
  - Research Site, Tonnoy, Lorraine
  - Research Site, Toul, Lorraine
  - Research Site, Vandœuvre-lès-Nancy, Lorraine
  - Research Site, Bron, Lyonnais
  - Research Site, Francheville, Lyonnais
  - Research Site, Gleizé, Lyonnais
  - Research Site, Lyon, Lyonnais
  - Research Site, Pont-Évêque, Lyonnais
  - Research Site, Ajaccio, Maures Corse
  - Research Site, Bormes-les-Mimosas, Maures Corse
  - Research Site, Furiani, Maures Corse
  - Research Site, Saint-Cyr-sur-Mer, Maures Corse
  - Research Site, Six-Fours-les-Plages, Maures Corse
  - Research Site, Toulon, Maures Corse
  - Research Site, Albi, Midi Pyrenees
  - Research Site, Blagnac, Midi Pyrenees
  - Research Site, Castanet-Tolosan, Midi Pyrenees
  - Research Site, La Tour-du-Crieu, Midi Pyrenees
  - Research Site, Lacrouzette, Midi Pyrenees
  - Research Site, Plaisance-du-Touch, Midi Pyrenees
  - Research Site, Toulouse, Midi Pyrenees
  - Research Site, Villeneuve-Tolosane, Midi Pyrenees
  - Research Site, Paris, Paris Centre
  - Research Site, Champs-sur-Marne, Paris Nord Est
  - Research Site, Gagny, Paris Nord Est
  - Research Site, Le Bourget, Paris Nord Est
  - Research Site, Lognes, Paris Nord Est
  - Research Site, Montfermeil, Paris Nord Est
  - Research Site, Angers, Pays de Loire
  - Research Site, Carquefou, Pays de Loire
  - Research Site, Champigné, Pays de Loire
  - Research Site, Cholet, Pays de Loire
  - Research Site, Nantes, Pays de Loire
  - Research Site, Saint-Laurent-de-la-Plaine, Pays de Loire
  - Research Site, Saint-Lyphard, Pays de Loire
  - Research Site, Saint-Nazaire, Pays de Loire
  - Research Site, Thouaré-sur-Loire, Pays de Loire
  - Research Site, Amiens, Picardie
  - Research Site, Le Quesnoy, Picardie
  - Research Site, Saint-Quentin, Picardie
  - Research Site, Wallers, Picardie
  - Research Site, Marignane, Provence-Alpes-Côte d'Azur Region
  - Research Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Miramas, Provence-Alpes-Côte d'Azur Region
  - Research Site, Fleury-les-Aubrais, Sologne
  - Research Site, Montigny-sur-Loing, Sologne
  - Research Site, Orléans, Sologne
  - Research Site, Vennecy, Sologne
  - Research Site, La Riche, Touraine
  - Research Site, Limeray, Touraine
  - Research Site, Tours, Touraine
  - Research Site, Dieulefit, Vallee Du Rhone
  - Research Site, Noves, Vallee Du Rhone
  - Research Site, Taillades, Vallee Du Rhone
  - Research Site, Beauvais, Vexin
  - Research Site, Cergy, Vexin
  - Research Site, Gonesse, Vexin
  - Research Site, Saint-Just-en-Chaussée, Vexin
  - Research Site, Vauréal, Vexin
  - Research Site, Argenteuil, Yvelines
  - Research Site, Élancourt, Yvelines
  - Research Site, Le Chesnay, Yvelines